CLINICAL TRIAL: NCT02480621
Title: The Impact of Liposomal Bupivicaine on Post-Operative Pain in Orthopaedic Trauma Surgery: A Double-Blind Prospective Randomized Control Trial
Brief Title: Liposomal Bupivacaine With Bupivacaine in Ankle Fracture Open Reduction Internal Fixation (ORIF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jamaica Hospital Medical Center (Other)
Responsible Party: Principal Investigator, Roy Davidovitch, M.D., Assistant Professor of Orthopaedic Surgery, Jamaica Hospital Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 623477-4
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Ankle Fracture
MeSH Terms: conditions — Ankle Fractures | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard of care: Open Reduction Internal Fixation with no injection of pain medications around the affected ankle.
- Liposomal Bupivacaine with Bupivacaine (Experimental): Intra-operatively, patients receive a local injection of liposomal bupivacaine with bupivacaine around the affected ankle.
  Interventions: Drug: Liposomal Bupivacaine with Bupivacaine

INTERVENTIONS:
Drug: Liposomal Bupivacaine with Bupivacaine — Pain medications injected locally during surgery around affected ankle.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine with Bupivacaine

SUMMARY:
This study is a randomized controlled trial assessing pain control in ankle fractures repaired with open reduction and internal fixation. Patients are consented and enrolled pre-operatively, and randomized to either control or liposomal bupivacaine with bupivacaine administered intra-operatively.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial assessing pain control in ankle fractures repaired with open reduction and internal fixation. Patients are consented and enrolled pre-operatively, and randomized to either control or liposomal bupivacaine with bupivacaine administered intra-operatively. Patients are to remain blinded to the treatment arm. The surgeon is non-blinded and administers the bupivacaine solution locally, intra-operatively.

Patients pain scores and pain medication usage is documented. A trained research coordinator contacts each patient at 24, 48, and 72 hours post-operatively to assess pain levels on a visual analog scale (VAS) and pain medications taken. Patients return for followup at standard intervals of 2 weeks, 6 weeks, 3 months, 6 months, and 1 year post-operatively to assess healing and functional outcomes. Patients are queried as to satisfaction with pain control at 2 weeks post-operatively. The study will compare outcomes including pain levels, pain medications taken, operating room (OR) and post-anesthesia care unit (PACU) times, length of stay (LOS), satisfaction with pain control, clinical outcomes, and complication rates.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years old.
2. Male or Female
3. All racial and ethnic groups
4. Fractures and fracture/dislocations of the ankle
5. Patients who opt for surgical treatment of their fractures.
6. Patients who consent to be randomized.
7. Patients who are willing to follow-up for a minimum of 52 weeks.

Exclusion Criteria:

1. Patients younger than 18 years old
2. Patients who are on chronic opioids
3. Patients who abuse opioids
4. Patients who are unwilling to follow-up for a minimum of 52 weeks
5. Neurologic condition that could interfere with pain sensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06-30 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Davidovitch, MD, Principal Investigator — Jamaica Hospital Medical Center
Locations (1):
- Jamaica Hospital Medical Center, Jamaica, New York, United States

REFERENCES:
- [Background] Owen RT. Bupivacaine liposome injectable suspension: a new approach to postsurgical pain. Drugs Today (Barc). 2013 Aug;49(8):475-82. doi: 10.1358/dot.2013.49.8.2006992. PMID 23977664
- [Background] Joshi GP, Cushner FD, Barrington JW, Lombardi AV Jr, Long WJ, Springer BD, Stulberg BN. Techniques for periarticular infiltration with liposomal bupivacaine for the management of pain after hip and knee arthroplasty: a consensus recommendation. J Surg Orthop Adv. 2015 Spring;24(1):27-35. PMID 25830260
- [Background] Lonner JH, Scuderi GR, Lieberman JR. Potential utility of liposome bupivacaine in orthopedic surgery. Am J Orthop (Belle Mead NJ). 2015 Mar;44(3):111-7. PMID 25750943
- [Background] Robbins J, Green CL, Parekh SG. Liposomal bupivacaine in forefoot surgery. Foot Ankle Int. 2015 May;36(5):503-7. doi: 10.1177/1071100714568664. Epub 2015 Jan 22. PMID 25614060

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Standard of care: Open Reduction Internal Fixation with no injection of pain medications around the affected ankle, but these control patients did receive a local intra-operative injection saline while under general anesthesia
Period: Randomization
Arm/Group | Control | Liposomal Bupivacaine With Bupivacaine
Started | 44 | 40
Completed | 43 | 39
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Surgeon did not give intervention | 0 | 1
Period: Follow Up
Arm/Group | Control | Liposomal Bupivacaine With Bupivacaine
Started | 43 | 39
Completed | 39 | 37
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Liposomal Bupivacaine With Bupivacaine | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 32 | 70
  >=65 years | 1 | 5 | 6
Age, Continuous [Mean (Full Range); unit: years] | 42.6 [19 to 69] | 41.9 [19 to 81] | 42 [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 20 | 18 | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 37 | 76
Body Mass Index (BMI) [Mean (Full Range); unit: kilogram per meter squared] | 29.7 [19.1 to 42] | 29.4 [17.9 to 48.1] | 29.5 [17.9 to 48.1]
Charlson Comorbidity Index (CCI) [Mean (Full Range); unit: units on a scale] — The CCI is a validated index used to quantitatively measure the number and severity of a patient's co-morbid illnesses. A specific grading chart for the various types and severity of illnesses is used that ranges from 0 points (i.e., no active disease process) to 6 points (i.e., most severe active disease process). Each illness is assigned a point value according to the scale, and the presence and severity of each illness are summed for an individual patient. A score of 0 indicates no active co-morbid illnesses within a patient, whereas a score >0 suggests 1 or more active disease processes.
  units on a scale | 0.9 [0 to 3] | 0.8 [0 to 5] | 0.88 [0 to 5]
OTA Fracture Classification [Count of Participants; unit: Participants] — The number of participants within each ankle fracture classification using the groupings provided by the Orthopaedic Trauma Association (OTA) (i.e., 44A, 44B, 44C) was determined. The numbering indicates the anatomic location of the fractures (i.e., 44 designates fractures of the tibia and/or fibula malleoli [ankle]). The lettering indicates the relative location of the fracture in regards to the location of the syndesmotic joint connecting the tibia and fibula such that A indicates fractures below this joint, B indicates fractures involving the joint, and C indicate fractures above the joint.
  Participants
    44A | 12 | 8 | 20
    44B | 16 | 19 | 35
    44C | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Pain Levels on a Visual Analog Scale ( VAS)
Description: A Visual Analog Scale (VAS) ranging from 0 to 10 in increments of 1 was used to both qualitatively and quantitatively assess the level and severity of pain during the time points ranging from the immediate post-operative period through 72 hours post-operative. Each number on the scale is accompanied by a visual facial expression that indicates the level of pain, discomfort, and distress appropriate to the number on the scale. The more severe the level of pain, the higher the corresponding number and more distressing the accompanying facial expression. A VAS score of 0 indicates no active pain level and is accompanied by a pleasantly smiling face whereas a VAS score of 10 indicates the most severe active pain level and is accompanied by a visibly-distraught face that is frowning, grimacing, and sweating. The combination of facial expressions and numbers is supposed to provide a language-independent, validated means of assessing pain levels.
Time Frame: Immediate post-operative period until 72 hours post-operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Liposomal Bupivacaine With Bupivacaine
Number analyzed (Participants) | 39 | 37
units on a scale
  4 Hours Post-operative | 7.05 (2.87) | 4.03 (3.50)
  Post-operative Day 1 | 7.49 (1.92) | 6.60 (1.85)
  Post-operative Day 2 | 6.64 (2.01) | 5.22 (1.81)
  Post-operative Day 3 | 5.72 (1.91) | 4.08 (1.85)
Statistical Analysis 1: Comparison: Control vs Liposomal Bupivacaine With Bupivacaine; Test type: Superiority; p < 0.10, t-test, 2 sided; Mean Difference (Net) = 1.74

ADVERSE EVENTS:
Time Frame: Patients were assessed for the development of any adverse events from the time of initial consent and enrollment through the their 6 month functional outcomes follow up.
Arm/Group | Control | Liposomal Bupivacaine With Bupivacaine
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/37
Other Adverse Events (participants affected / at risk) | 0/39 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No